CLINICAL TRIAL: NCT05273957
Title: A Model of Hospital-territory Management Coordinated by a Case Manager to Improve the Care of Patients With Parkinsonism. A Multicenter, Randomized, Double-blind Study. The PROUD Study
Brief Title: A Model of Hospital-Territory Management Coordinated by a Case Manager to Improve the Care of Patients With Parkinsonism.
Acronym: PROUD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Azienda Socio Sanitaria Territoriale Nord Milano (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PROUD
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease; Atypical Parkinsonism; Secondary Parkinsonism; Nurse-Patient Relations; Nurse Physician Relations
Keywords: Parkinson Disease; Case Manager; Parkinson Disease Nurse Specialist
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease, Secondary | interventions — Case Managers; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Manager (Experimental): Patients are followed up by a case manager
  Interventions: Other: Case Manager
- Standard-of-care (Active Comparator): Patients are followed up only by the neurologist
  Interventions: Other: Standard-of-care

INTERVENTIONS:
Other: Case Manager — Patients are followed up by a nurse specialist in parkinsonism (case manager) who interacts with the treating neurologist and a multidisciplinary team
  Arms: Case Manager
Other: Standard-of-care — Patients are managed only by the neurologist according the institution's clinical practice
  Arms: Standard-of-care

SUMMARY:
The present multicenter randomized study investigates whether the management of patients with parkinsonism by a nurse specialist (case-manager) can significantly improve patients' quality of life over 12 months, compared to control patients managed with the standard-of-care process.

Participants will be evaluated with clinical scales testing quality of life, motor and non-motor symptoms, and the number of unscheduled hospital access throughout the course of the study.

DETAILED DESCRIPTION:
Several studies provide evidence that a multidisciplinary management of individuals with Parkinson's disease (PD) including a specialized nurse may offer significant benefits to patients, in the management of disability due to motor and non-motor symptoms as well as in monitoring compliance to therapy and incident adverse events.

A number of retrospective studies demonstrated that frequent neurologic consultations and a strict adherence to pharmacological therapy can reduce the risk of hospitalization up to 50%. Falls, fractures, infections and cognitive and motor deterioration represent risk factors for hospitalization in patients with PD. These complications are even more frequent in patients affected by atypical parkinsonisms (e.g. multiple system atrophy and progressive supranuclear palsy).

The optimization of management of motor and non-motor symptoms and pharmacological side effects, through telemedicine services carried out by nurses specialized in movement disorders, can prevent falls and hospitalization, increase quality of life and reduce comorbidities and caregiver's burnout.

In the present study, a "case-manager" will follow-up patients and caregivers, cooperating at the same time with other members of a multidisciplinary team (neurologists, psychologists, physiatrists, general practitioners, social assistants), either within or outside the institute where the neurologist visits, aiming to achieve a better global management of frail patients.

The present multicenter, randomized, double-blind study will recruit 164 patients affected by Parkinson's disease, atypical parkinsonism or secondary parkinsonism with motor and/or non motor complications, living in the Lombardy region (Northern Italy).

Patients will be enrolled in a tertiary referral clinic with expert knowledge ('hub': Fondazione IRCCS Istituto Neurologico Carlo besta) and in a community hospital ('spoke': Azienda Socio Sanitaria Territoriale Nord Milano).

The participants will be randomized into two treatment arms: (i) the interventional arm (patients followed by a case manager); (ii) the control arm (the standard-of-care).

At the baseline and at the visits at 6 and 12 months, clinical scales and questionnaires will be administered to determine if there are differences between the quality of life and the disability of patients between the two arms of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Living in the Lombardy region (Northern Italy)
* Duration of Parkinson's disease, atypical or secondary parkinsonism ≥ 3 years
* Presence of at least (i) n=1 motor complication and/or (ii), n=2 non-motor symptoms, defined as follows:

  (i) Motor complication:
* Motor fluctuations
* ≥ 2 Falls in the last 6 months
* Dysphagia

(ii) Non Motor symptoms

* Non-motor fluctuations
* ≥ 2 items of the non-motor symptoms scale with a score ≥ 2

Exclusion Criteria:

* Hoehn and Yahr Stage = 5 in the ON-medication condition
* Psychiatric comorbidity or other neurological chronic diseases that, in the opinion of the recruiting neurologist, could compromise the study participation.
* Patients on infusional therapies (continuous infusion of levodopa-carbidopa intestinal gel or Continuous Subcutaneous Apomorphine Infusion).
* Severe medical disease (liver or kidney failure, decompensated heart disease, neoplasms, coagulopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in total score of the Parkinson's Disease Questionnaire 39-items scale | baseline, week 52
  Thi is a 39-items questionnaire assessing the quality of life of patient with Parkinson's disease. The higher the score the lower the quality of life

SECONDARY OUTCOMES:
Number of unscheduled hospital access over the 12-month study period | baseline, week 26, week 52
  The investigators will collect the sum of the number of (i) extra unscheduled outpatient visits, (ii) emergency room visits, (iii) hospital admissions directly or indirectly associated with parkinsonism
Changes in the Movement Disorder Society Unified Parkinson's Disease Rating Scale part II | baseline, week 52
  This is a scale (MDS-UPDRS) used to assess activities of daily living. The higher the score the worse the Disability
Changes in the Movement Disorder Society Unified Parkinson's Disease Rating Scale part IV | baseline, week 52
  This is a scale (MDS-UPDRS) used to assess complications of dopaminergic therapy. The higher the score the worse the disability
Changes in the Non-Motor Symptoms Scale score | baseline, week 52
  This is a scale used to assess the burden of non-motor symptoms in Parkinson's disease. The higher the score the worse the disability
Changes in the activities of daily living questionnaire | baseline, week 52
  The "ADL (Activities of Daily Living)" evaluation refers to the fundamental activities of daily life in which the subject is dependent: on a scale from 0 to 6 points, the lower the score, the greater the person's need for assistance
Changes in the instrumental activities of daily living questionnaire | baseline, week 52
  The "IADL (Instrumental Activities of Daily Living)" evaluation refers to the instrumental activities of daily life in which the subject is dependent (eg using telephone, preparing meals, taking medications, etc): on a scale from 0 to 8 points, the lower the score, the greater the person's need for assistance
Changes in patient experience questionnaire | baseline, week 26, week 52
  This is a questionnaire assessing patient perception and satisfaction of the quality of health care
Changes in EuroQOL-5 Dimensions-5 Levels score | baseline, week 52
  This is a useful and validated instrument to measure quality of life in patients with Parkinson's disease
Changes in the Morisky Medical Adherence scale-8 items score | baseline, week 26, week 52
  This is an 8-items scale used to investigate patient adherence to the therapy prescribed by the MD specialist
Changes in the Zarit Burden Interview scale score | baseline, week 26, week 52
  This is a scale used to investigate caregiver's burnout
Number of incident comorbidities | baseline, week 26, week 52
  The number of incident comorbidities over the 12.month study period will be assessed using a semistructured interview

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Eleopra, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (2):
- Italy (2):
  - Azienda Socio-Sanitaria Territoriale Nord Milano, Sesto San Giovanni, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest on this topic. Data shared will be coded, with no protected health information included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months.
  Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement. For more information or to submit a request, please contact crc@istituto-besta.it

REFERENCES:
- [Background] van der Marck MA, Bloem BR, Borm GF, Overeem S, Munneke M, Guttman M. Effectiveness of multidisciplinary care for Parkinson's disease: a randomized, controlled trial. Mov Disord. 2013 May;28(5):605-11. doi: 10.1002/mds.25194. Epub 2012 Nov 19. PMID 23165981
- [Background] Willis AW, Schootman M, Tran R, Kung N, Evanoff BA, Perlmutter JS, Racette BA. Neurologist-associated reduction in PD-related hospitalizations and health care expenditures. Neurology. 2012 Oct 23;79(17):1774-80. doi: 10.1212/WNL.0b013e3182703f92. Epub 2012 Oct 10. PMID 23054239
- [Background] Muzerengi S, Herd C, Rick C, Clarke CE. A systematic review of interventions to reduce hospitalisation in Parkinson's disease. Parkinsonism Relat Disord. 2016 Mar;24:3-7. doi: 10.1016/j.parkreldis.2016.01.011. Epub 2016 Jan 13. PMID 26803377
- [Background] Gerlach OH, Broen MP, van Domburg PH, Vermeij AJ, Weber WE. Deterioration of Parkinson's disease during hospitalization: survey of 684 patients. BMC Neurol. 2012 Mar 8;12:13. doi: 10.1186/1471-2377-12-13. PMID 22400982
- [Background] Hassan A, Wu SS, Schmidt P, Dai Y, Simuni T, Giladi N, Bloem BR, Malaty IA, Okun MS; NPF-QII Investigators. High rates and the risk factors for emergency room visits and hospitalization in Parkinson's disease. Parkinsonism Relat Disord. 2013 Nov;19(11):949-54. doi: 10.1016/j.parkreldis.2013.06.006. Epub 2013 Jul 5. PMID 23835430
- [Background] Low V, Ben-Shlomo Y, Coward E, Fletcher S, Walker R, Clarke CE. Measuring the burden and mortality of hospitalisation in Parkinson's disease: A cross-sectional analysis of the English Hospital Episodes Statistics database 2009-2013. Parkinsonism Relat Disord. 2015 May;21(5):449-54. doi: 10.1016/j.parkreldis.2015.01.017. Epub 2015 Feb 17. PMID 25737205
- [Background] Peto V, Jenkinson C, Fitzpatrick R. PDQ-39: a review of the development, validation and application of a Parkinson's disease quality of life questionnaire and its associated measures. J Neurol. 1998 May;245 Suppl 1:S10-4. doi: 10.1007/pl00007730. PMID 9617716
- [Background] Schrag A, Selai C, Jahanshahi M, Quinn NP. The EQ-5D--a generic quality of life measure-is a useful instrument to measure quality of life in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2000 Jul;69(1):67-73. doi: 10.1136/jnnp.69.1.67. PMID 10864606
- [Background] Hellqvist C, Bertero C. Support supplied by Parkinson's disease specialist nurses to Parkinson's disease patients and their spouses. Appl Nurs Res. 2015 May;28(2):86-91. doi: 10.1016/j.apnr.2014.12.008. Epub 2015 Feb 26. PMID 25908544
- [Background] van der Eijk M, Faber MJ, Ummels I, Aarts JW, Munneke M, Bloem BR. Patient-centeredness in PD care: development and validation of a patient experience questionnaire. Parkinsonism Relat Disord. 2012 Nov;18(9):1011-6. doi: 10.1016/j.parkreldis.2012.05.017. Epub 2012 Jun 15. PMID 22704902
- [Background] Qiang JK, Marras C. Telemedicine in Parkinson's disease: A patient perspective at a tertiary care centre. Parkinsonism Relat Disord. 2015 May;21(5):525-8. doi: 10.1016/j.parkreldis.2015.02.018. Epub 2015 Feb 28. PMID 25791380
- [Background] Hagell P, Alvariza A, Westergren A, Arestedt K. Assessment of Burden Among Family Caregivers of People With Parkinson's Disease Using the Zarit Burden Interview. J Pain Symptom Manage. 2017 Feb;53(2):272-278. doi: 10.1016/j.jpainsymman.2016.09.007. Epub 2016 Nov 1. PMID 27810571
- [Background] Cova I, Di Battista ME, Vanacore N, Papi CP, Alampi G, Rubino A, Valente M, Meco G, Contri P, Di Pucchio A, Lacorte E, Priori A, Mariani C, Pomati S. Validation of the Italian version of the Non Motor Symptoms Scale for Parkinson's disease. Parkinsonism Relat Disord. 2017 Jan;34:38-42. doi: 10.1016/j.parkreldis.2016.10.020. Epub 2016 Oct 24. PMID 28029554
- [Background] Fabbrini G, Abbruzzese G, Barone P, Antonini A, Tinazzi M, Castegnaro G, Rizzoli S, Morisky DE, Lessi P, Ceravolo R; REASON study group. Adherence to anti-Parkinson drug therapy in the "REASON" sample of Italian patients with Parkinson's disease: the linguistic validation of the Italian version of the "Morisky Medical Adherence Scale-8 items". Neurol Sci. 2013 Nov;34(11):2015-22. doi: 10.1007/s10072-013-1438-1. Epub 2013 Jun 1. PMID 23728715
- [Background] Bloem BR, Henderson EJ, Dorsey ER, Okun MS, Okubadejo N, Chan P, Andrejack J, Darweesh SKL, Munneke M. Integrated and patient-centred management of Parkinson's disease: a network model for reshaping chronic neurological care. Lancet Neurol. 2020 Jul;19(7):623-634. doi: 10.1016/S1474-4422(20)30064-8. Epub 2020 May 25. PMID 32464101
- [Background] Cilia R, Mancini F, Bloem BR, Eleopra R. Telemedicine for parkinsonism: A two-step model based on the COVID-19 experience in Milan, Italy. Parkinsonism Relat Disord. 2020 Jun;75:130-132. doi: 10.1016/j.parkreldis.2020.05.038. Epub 2020 Jun 10. PMID 32723588